CLINICAL TRIAL: NCT04442932
Title: Validation of the abioSCOPE Device With an IgE Test Panel: Clinical Sensitivity and Specificity Study
Brief Title: abioSCOPE IgE Assay to Aid in the Diagnosis of Allergies
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor financial has been stopped.
Sponsor: Abionic SA (Industry)
Collaborators: NAMSA (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: AB-ALL-003.2
Record Dates: First submitted 2020-06-16; First posted 2020-06-23 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Allergy; Allergic Asthma; Allergy to Cats; Allergy to House Dust; Allergy to Dog Dander; Allergy Cockroach
Keywords: Allergy; Asthma; Point-of-Care; Immunoassay; In vitro Diagnostic; Total IgE; Specific allergy
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Interventions: Per test, a minimum of 40 atopic subjects for a given allergy and a total of at least 100 non-atopic subjects. To ensure that sufficient subjects with valid results are enrolled, the atopic enrollment goal per allergy is approximately 50 subjects. For each allergen, approximately 20% of the samples must be in the range of 0.70 to 3.5 IUA/mL and the remainder must cover a measuring range that is representative of the target population. Results from a single positive subject can be used in the analyses of more than one allergen if the subject is sensitized for more than one allergen.
  Interventions: Device: Blood Collection

INTERVENTIONS:
Device: Blood Collection — K3-EDTA venous whole blood 9 mL 1 venous draw

SUMMARY:
This is a multicenter, prospective, observational study designed to determine the clinical sensitivity and specificity of the Abionic IVD CAPSULE Allergic Asthma panel performed on Abionic's abioSCOPE device using K3-EDTA anticoagulated plasma samples from atopic and non-atopic pediatric and adult patients. Patients' sensitization determined with the abioSCOPE will be compared to the clinical assessment of allergy.

ELIGIBILITY:
Inclusion Criteria:

Atopic and non-atopic individuals are needed for this study. For enrollment in the atopic arm, patients must meet all of the inclusion criteria listed below to be eligible for participation:

1. Provide signed and dated written informed consent by patient or legally designated representative prior to any mandatory study-specific procedures, sample collection, or analysis. Assent will be obtained from pediatric patients who are ≥ 6 years of age and less than 18 years of age.
2. Male or female, ≥ 6 years of age.
3. Consulting for signs and/or symptoms of IgE-mediated allergies to perennial allergens.

For enrollment in the non-atopic arm, patients must meet all of the inclusion criteria list below to be eligible for participation:

1. Provide signed and dated written informed consent by patient or legally designated representative prior to any mandatory study-specific procedures, sample collection, or analysis. Assent will be obtained from pediatric patients who are ≥ 6 years of age and less than 18 years of age.
2. Male or female, ≥ 6 years of age.
3. Apparently healthy individuals who exhibit no signs/symptoms of IgE-mediated allergies including rhinitis, conjunctivitis, asthma, eczema, urticaria or food allergy symptoms upon exposure to animal danders, dust mites, cockroaches, pollens or food allergens (non-atopic).

Exclusion Criteria:

Patients must not meet any exclusion criteria below to be eligible for participation:

1. Patient participating in another study that may influence test results.
2. Subjects taking any of the following medications: antihistamines in the week preceding the consultation, systemic steroids (inhaled or nasal steroids are allowed), anti-cytokines or cytokines, systemic interferon (injection local interferon α for the treatment of HPV is allowed), anti-IgE therapy (approved or investigational) or treated with systemic chemotherapy.
3. On-going allergen immunotherapy or prior allergen immunotherapy within the prior 3 years.
4. Patient with a history of cancer, autoimmune, or immune deficiency disease.
5. Patient suffering from a hematological pathology (coagulation disorder, severe anemia) that could interfere with the blood test.
6. Known severe allergic reaction to any of the IVD CAPSULE Allergic Asthma panel allergen components

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: • Per test, a minimum of 40 atopic subjects for a given allergy and a total of at least 100 non-atopic subjects (). To ensure that sufficient subjects with valid results are enrolled, the atopic enrollment goal per allergy is approximately 50 subjects. For each allergen, approximately 20% of the samples must be in the range of 0.70 to 3.5 IUA/mL and the remainder must cover a measuring range that is representative of the target population. Results from a single positive subject can be used in the analyses of more than one allergen if the subject is sensitized for more than one allergen.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the abioSCOPE | Day 1
  The primary objective will be evaluated by estimating the Sensitivity and Specificity of the abioSCOPE to detect sensitization to each of the five allergens or group of allergens. The estimates will be accompanied by 95% Clopper-Pearson Confidence Intervals. The acceptance criteria will be compared to the lower bound of the 95% confidence interval. The ability of the abioSCOPE to detect sensitization to each allergen will be considered acceptable if both the sensitivity and specificity of the allergen meet both performance goals.

OTHER OUTCOMES:
Determination of Positive Predictive Value (PPV), Negative Predictive Value (NPV), Concordance and study prevalence of allergen sensitization. | Day 1
  Presentation of Positive Predictive Value (PPV), Negative Predictive Value (NPV), Concordance and study prevalence of allergen sensitization based of the classification of 40 subjects for each allergen.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - George Washington University, Washington DC, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Creticos Research Group, LLC, Crownsville, Maryland
  - The Bernstein Clinical Research Center Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided